CLINICAL TRIAL: NCT03197155
Title: Direct-acting Antiviral Therapy Decreases Hepatocellular Carcinoma Recurrence Rate in Cirrhotic Patients With Chronic Hepatitis C
Brief Title: Direct-acting Antivirals and Hepatocellular Carcinoma Recurrence
Acronym: RECAR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0400
Record Dates: First submitted 2017-06-12; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Hepatocellular Carcinoma; Hepatitis C; Direct Acting Antivirals
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Direct Acting Antivirals against hepatitis C virus infection — The cohort includes cirrhotic patients infected with HCV and successfully treated for their first history of hepatocellular carcinoma. Some of these patients were treated with direct-acting antivirals for their HCV infection while the others did not receive any direct-acting antivirals treatment during the follow-up period.

SUMMARY:
Background and Aims: Arrival of direct-acting antiviral (DAA) agents against hepatitis C virus (HCV) with high-sustained virological response (SVR) rates and very few side effects has drastically changed the management of HCV infection. The impact of DAA exposure on hepatocellular carcinoma (HCC) recurrence after a first remission in patients with advanced fibrosis remains to be clarified.

Methods: 68 consecutive HCV patients with a first HCC diagnosis and under remission, subsequently treated or not with a DAA combination, were included. Clinical, biological, and virological data were collected at first HCC diagnosis, at remission and during the surveillance period.

ELIGIBILITY:
Inclusion Criteria:

* first HCC diagnosed by invasive or non-invasive criteria following the American Association for the Study of Liver Diseases (AASLD) guidelines during the study time horizon
* complete remission after hepatocellular carcinoma treatment defined by the European Association for the Study of the Liver (EASL) criteria as absence of residual tumor/complete necrosis at imaging one month after the end of hepatocellular carcinoma treatment

Exclusion Criteria:

* prior history of hepatocellular carcinoma before January 2009
* liver transplantation before hepatocellular carcinoma diagnosis
* presence of "non-characterized nodules" after hepatocellular carcinoma treatment at imaging
* history of direct-acting antivirals treatment before the first hepatocellular carcinoma diagnosis
* hepatic decompensation
* human immunodeficiency virus (HIV) coinfection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HCV infected patients from the Department of Hepatology, Croix-Rousse Hospital, Lyon, France developing a first HCC and receiving or not a direct-acting antiviral combination therapy after HCC remission between January 2009 and March 2016 were considered.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Hepatocellular recurrence event | From date of HCC remission until the date of HCC recurrence, assessed up to January 1st, 2017
  The primary outcome (hepatocellular recurrence event) is evaluated using imaging surveillance data at different time points during follow-up (every 3 months within the first year following HCC remission and every 3 to 6 months thereafter) after the first HCC remission.

IPD SHARING:
Plan to Share IPD: No